CLINICAL TRIAL: NCT03702803
Title: Efficacy and Safety Study of a IMSS Developed Phytopharmaceutical for the Treatment of Anxiety. Double Blind and Randomized Clinical Trial Controlled With Alprazolam
Brief Title: Efficacy and Safety Study of a IMSS Developed Phytopharmaceutical for the Treatment of Anxiety.
Acronym: Alpra
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Jaime Tortoriello García, Head of Southern Biomedical Research Center, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Galphimia glauca phytopharm
Record Dates: First submitted 2018-10-01; First posted 2018-10-11 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Phytopharmaceutical; Anxiety; Outpatients
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two groups: the experimental group receiving a phytopharmaceutical elaborated with the standardized extract from G. glauca, and a control group receiving an identical formulation containing Alprazolam
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both treatments have an identical appearance and are packed in hard gelatin capsules, which are packed in individual aluminum and PVC blisters with 10 doses each. Three blisters with ten doses are introduced in cardboard boxes and identified through a folio number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galphimia glauca standardized extract (Experimental): Patients with a clinical diagnosis of GAD (with a score of 18 points or more on the Hamilton anxiety scale) that will be included in the experimental group and will be assigned the treatment consisting of hard gelatin capsules with a pharmaceutical formulation prepared with a standardized extract from G. glauca, which will be administered once a day.
  Interventions: Dietary Supplement: Galphimia glauca standardized extract
- alprazolam 1mg (Active Comparator): Patients with a clinical diagnosis of GAD (with a score of 18 points or more on the Hamilton anxiety scale) that will be included in the control group and will be assigned the treatment consisting of hard gelatin capsules with the drug Alprazolam (1 mg ), which will be administered once a day.
  Interventions: Drug: alprazolam 1mg

INTERVENTIONS:
Dietary Supplement: Galphimia glauca standardized extract — Each patient will be administered with a capsule once a day (in the morning), for 10 weeks. A capsule contains the standardized extract of Galphimia glauca corresponding to 0.374 mg of Galphimine-B
  Arms: Galphimia glauca standardized extract
Drug: alprazolam 1mg — Each patient will be administered once a day (in the morning) for 10 weeks. A capsule contains 1 mg Alprazolam
  Other Names: Alprazolam
  Arms: alprazolam 1mg

SUMMARY:
The investigator's group at the Mexican Institute of Social Security has worked for more than 20 years in the scientific research of the plant species Galphimia glauca Cav., which is used in Mexican Traditional Medicine for the treatment of mental disorders. With the obtained results it was possible the development of a phytopharmaceutical elaborated with the extract of this plant, which was standardized in its content of Galphimine-B (G-B). This new compound is a nor, seco-triterpene, which possesses selective effects on the central nervous system. Through electrophysiological neuronal unitary records it was identified that G-B acts on the ventral tegmental area (VTA), and exerts its effect on (N-methyl-D-aspartate) NMDA receptors in dopaminergic neurons. The new phytopharmaceutical, elaborated from a standardized extract (in its G-B content) of G. glauca, was subjected to a double blind and randomized clinical study that compared its efficacy and therapeutic tolerability with a similar drug formulated with lorazepam in patients with diagnosis of generalized anxiety disorder (GAD). In a total of 152 patients, it was evidenced that the phytomedicine administered orally (for 4 weeks) was able to significantly reduce anxiety, in a similar way as lorazepam did, but with better tolerability. Several patients who were treated with lorazepam had to leave the study because they had daytime sleepiness.

In clinical practice, different benzodiazepines have specific indications. In the case of anxiety disorders, the drug of first choice is Alprazolam, this, because it manifests a more powerful anxiolytic effect with a lower degree of sedation and daytime sleepiness.

Objective: The present project aims to compare the efficacy and therapeutic safety of an elaborated phytopharmaceutical with the standardized extract of Galphimia glauca with Alprazolam .

DETAILED DESCRIPTION:
A double-blind, randomized, controlled clinical study will be conducted in patients with GAD.

The development of the phytopharmaceutical will be carried out at the Southern Biomedical Research Center, belonging to the Mexican Institute of Social Security. The preparation of the plant material, extraction, concentration, standardization of the vegetable drug, the design and production of the experimental drug as well as the control treatment will be carried out in this site.

The clinical trial will be developed with outpatient from the Primary Care Family Medicine Unit of the Regional General Hospital No. 1 of the Mexican Institute of Social Security in Cuernavaca, Morelos, Mexico.

SUBJECTS. Patients of both sexes aged 18 years and older who present Generalized Anxiety disorder (GAD) and who meet the selection criteria.

Experimental group Patients with a clinical diagnosis of GAD (with a score of 18 points or more on the Hamilton anxiety scale) that will be included in the experimental group and will be assigned the treatment consisting of hard gelatin capsules with a pharmaceutical formulation prepared with a standardized extract (in its content of Galphimine-B, G-B) of G. glauca, which will be administered once a day.

Control group Patients with a clinical diagnosis of GAD (with a score of 18 points or more on the Hamilton anxiety scale) that will be included in the control group and will be assigned the treatment consisting of hard gelatin capsules with the drug Alprazolam (1 mg ), which will be administered once a day.

GENERAL DESCRIPTION OF THE STUDY The project will be promoted through posters that will be placed in strategic areas of the Medical Unit. In addition, brochures will be distributed with information about anxiety and the requirements to enter the project. There will also be support staff, Who will be in charge of giving conferences related with GAD in the waiting Hospital rooms. Once a person is identified who is a candidate to be included in the study, an invitation will be made to go to the clinical research office for evaluation.

In the research office, a trained physician, will practice the candidates a medical history and physical examination. The above, with the purpose of corroborating the diagnosis of GAD through the application of the Hamilton Anxiety Scale. This fully validated instrument will serve to make the clinical diagnosis of the condition.

If the questionnaire applied to the candidate gives us a total score of 18 points or more, the patient will be considered a candidate to enter the study. In order to be admitted, the patient, in addition must to have a clinical diagnosis of GAD, must meet the selection criteria established in this study. Once the patient complies with these two aspects will be given the necessary information about the study and about their participation in it. Patient must also sign a letter of informed consent, this letter will contain information about the characteristics of the study, benefits to the population, commitment that the patient acquires when participating, commitments that the researcher acquires when the patient is included and the rights that the participant acquires.

Each of the participants will be randomly assigned the corresponding medication (which can be experimental or control) through a procedure based on a table of random numbers. The dosage of medications will be every 24 hours, administered orally in the morning. The indication will be given that the medication is taken together with the food. The duration of the administration of the medication will be for ten weeks.

In addition, each of the patients will be provided oral and written instructions on the form and times to take the medication, as well as the possible adverse effects and hygienic-dietetic measures that must be taken.

The patient will be following weekly, but may go to receive care at the time you require it. At each appointment, the state of health and the evolution of the condition will be evaluated, and the overall improvement scale will also be applied. At each appointment, patient will be given a control card (to each patient) where he will write down the days the medication was taken and whether or not there were any adverse effects during that administration period. In this way, adherence to treatment and tolerability will be evaluated.

The values of the Hamilton anxiety scale and the global improvement scale will be used to define the effectiveness, the therapeutic success or failure.

The final assessment of efficacy, tolerability, attachment and therapeutic success will be made during the last appointment. A summary will be sent to the family doctor of each of the participants and their discharge from the study.

SAMPLE SIZE The size of the sample was calculated according to the formula for comparison of two proportions, taking as background the efficacy that the species showed in previous clinical studies on generalized anxiety. The procedure yielded a total of 105 patients. 15% will be added to the sample size to compensate for possible losses, which leaves us with a final sample size of 122 patients.

DATA ANALYSIS. The results will be analyzed through descriptive statistics with frequencies and percentages. The X2 test will be used for the analysis of differences in proportions and ANOVA for mean differences, as well as Tukey's test for the difference between groups. Values of p less than 0.05 will be used to define differences between statistically significant groups

ETHICAL ASPECTS Project research was evaluated and approved by the National Scientific National Committee.

The species G. glauca has been used for many years in traditional Mexican medicine to treat some mental disorders. A pharmaceutical formulation, elaborated with the extract obtained from G. Glauca has been used in clinical projects to evaluate its efficacy and tolerability in patients with anxiety disorder. The administration time has been four weeks with a daily dose of a standardized product in 0.374 mg of G-B per dose. No significant adverse effects have been identified. Because it is a phytopharmaceutical that has shown good tolerability, the risk of adverse effects is low.

In developing this project, the aim is to have a novel alterative treatment that expresses a different mechanism of action, and that shows efficacy and tolerability in the treatment of GAD, but also that the effect obtained is comparable or better than that of a drug, elaborated with Alprazolam, which is the benzodiazepine of first choice and with specific indication for the treatment of this condition.

According to the Regulation of the General Law of Health in Research, there is no risk in the patients who will participate in the present project. The project will only include adults; will not include women with pregnancy or lactation or another sector vulnerable to research.

The research procedures are in accordance with the ethical rules of investigation, the Regulation of the General Law of Health in the field of health research and the Declaration of Helsinki and its amendments. All information obtained by conducting this study will be handled in a scientific and confidential manner. The clinical files will be kept under guard and the management of the information for the analysis of results will be done exclusively with the assigned folio number. No patient will be included if it is not widely known in which it will consist of their participation, the background of the medication, time that will last the study, dose that will be administered and frequency of the same, laboratory studies to which you will be subjected in addition to informing you that you have the freedom to withdraw from the study at the time you want. The patient will receive extensive and clear information about the protocol, the content of the letter of informed consent will be read, will be given space for the formulation of questions or concerns.

ASPECTS OF SECURITY The patients included in the study will be evaluated clinically in each of the appointments. In addition, at the beginning of the study and at the end of the administration period, laboratory tests will be performed to assess liver and kidney function. Medical surveillance with the search for adverse events will be included in each of the visits. In case of identifying any adverse effect, it will be monitored until its disappearance and the measures described below will be applied according to the event's rating.

An adverse event will be considered as any unpleasant, unintentional harmful medical occurrence that a patient submits to the administration of a pharmaceutical product, which may or may not have a causal relationship to the treatment.

The intensity of the adverse events refers to the maximum intensity with which the patient and / or the investigator qualify the adverse events that the patient presents.

1. Mild: The adverse effect is presented, but it is easily tolerated and does not require treatment
2. Moderate: the adverse effect is enough to interfere with normal activities
3. Severe: The adverse effect incapacitates the subject
4. Serious: Any adverse effect that results in the death of the patient, endangers life, requires hospitalization, causes disability or persistent or significant disability, causes a congenital anomaly or cancer, requiring surgical intervention to prevent permanent sequel or develop drug dependence or abuse Overdose is defined as the exposure without a specific therapeutic goal to an amount of medication of at least twice the maximum daily dose reported in the study protocol.

In all cases in which a severe adverse effect is identified, the treatment will be suspended and the patient will be removed from the study. In addition to the above, the patient will be referred for care in the specialized medical area and will be monitored until the resolution of the adverse effect. In the event of a serious adverse effect, the treatment will be suspended, the patient will be removed from the study and the blind code of the patient will be opened. In those cases in which there is a mild or moderate adverse effect, it will be reported in the patient's clinical file, it will be attended immediately and surveillance will be maintained until its complete remission. In these cases, the treatment will not be suspended, and the patient will remain within the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Eighteen years of age and older
* Clinical diagnosis of Generalized Anxiety Disorder
* Eighteen points or more on Hamilton Anxiety Scale
* Without previous treatment for this disease (for at least one month before).
* In case of being women of reproductive age, who are not pregnant or lactating.
* To sign an informed consent letter of participation in the investigation.

Exclusion Criteria:

* Patients who have treatment for their condition
* Patients who have another mental disorder added
* Patients with alcoholism, smoking or drug addiction
* Patients who live alone
* Ingest of drugs for insomnia
* Ingest of drugs of the Monoamine Oxidase Inhibitors group
* Patients with epilepsy
* Patients who operate dangerous machinery
* Patients who have to drive at work (car, truck or other motor vehicle) for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2020-09-19 (Estimated); Study Completion 2020-10-19 (Estimated)

PRIMARY OUTCOMES:
Therapeutic efficacy: improvement of the clinical condition higher than 90%. It will be measured by means of the Hamilton Rating Scale for Anxiety. | Up to 10 weeks
  It will be considered when the patient presents an improvement of the clinical condition higher than 90% on the scales of measurement (HAM-A). Hamilton Rating Scale for Anxiety (HAM-A) consisted of 14 items that assessed the severity of anxiety. Each item was scored using a 5-point scale (0=not present to 4=very severe). The HAM-A Total Score could have ranged from 0 to 56 and higher scores indicated a greater degree of symptom severity. Scores 14-21 indicate mild anxiety; scores 21-29 indicate moderate anxiety; scores over 29 indicate severe anxiety

SECONDARY OUTCOMES:
Therapeutic Tolerability: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 10 weeks
  Incidence and duration of adverse events monitored throughout the study by physical examination and the application of a questionnaire. It will by considered as Treatment Tolerability when the participant does not present adverse effect of Grade 3 according to the Common Terminology Criteria for Adverse Events v4.0
Clinical Global Impression of Improvement Scale (CGI-I). A 7 points scale that is used to evaluate how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. | Up to 10 weeks
  Clinical Global Impression of Improvement Scale is useful to evaluate the clinician's perception of the participant improvement at the time of assessment compared with the baseline condition, before initiating the intervention. The scale could have ranged from 1 to 7, where 1 means very much improved since the initiation of treatment; 2 means much improved; 3 means minimal improved; 4 means no change from baseline; 5 means minimally worse; 6 means much worse; 7 means very much worse.
  Values near to 1 or equal to 1 are considered better outcome, while higher values near to 7 or equal to 7 are considered worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: JAIME TORTORIELLO, Dr, Principal Investigator — Centro de Investigación Biomédica del Sur (CIBIS), IMSS; SUSANA NAVARRETE, DR, Study Chair — CIS MEXICO
Locations (1):
- Regional General Hospital Number 1 at Cuernavaca, Morelos. Mexican Insitute of Social Security, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plant to share IPD

REFERENCES:
- [Result] Tortoriello J, Lozoya X. Effect of Galphimia glauca methanolic extract on neuropharmacological tests. Planta Med. 1992 Jun;58(3):234-6. doi: 10.1055/s-2006-961442. PMID 1409977
- [Result] Tortoriello J, Ortega A. Sedative effect of galphimine B, a nor-seco-triterpenoid from Galphimia glauca. Planta Med. 1993 Oct;59(5):398-400. doi: 10.1055/s-2006-959717. PMID 8255929
- [Result] Tortoriello J, Ortega A, Herrera-Ruiz M, Trujillo J, Reyes-Vazquez C. Galphimine-B modifies electrical activity of ventral tegmental area neurons in rats. Planta Med. 1998 May;64(4):309-13. doi: 10.1055/s-2006-957440. PMID 9619110
- [Result] Osuna L, Pereda-Miranda R, Tortoriello J, Villarreal ML. Production of the sedative triterpene galphimine B in Galphimia glauca tissue culture. Planta Med. 1999 Mar;65(2):149-52. doi: 10.1055/s-1999-14057. PMID 10193207
- [Result] Prieto-Gomez B, Tortoriello J, Vazquez-Alvarez A, Reyes-Vazquez C. Galphimine B modulates synaptic transmission on dopaminergic ventral tegmental area neurons. Planta Med. 2003 Jan;69(1):38-43. doi: 10.1055/s-2003-37043. PMID 12567277
- [Result] Gonzalez-Cortazar M, Tortoriello J, Alvarez L. Norsecofriedelanes as spasmolytics, advances of structure-activity relationships. Planta Med. 2005 Aug;71(8):711-6. doi: 10.1055/s-2005-871224. PMID 16142633
- [Result] Rojas G, Aranda E, Navarro V, Zamilpa A, Tortoriello J. In vitro propagation of Galphimia glauca and content of the sedative compound galphimine-B in wild and micropropagated plants. Planta Med. 2005 Nov;71(11):1076-8. doi: 10.1055/s-2005-873136. PMID 16320215
- [Result] Herrera-Ruiz M, Jimenez-Ferrer JE, De Lima TC, Aviles-Montes D, Perez-Garcia D, Gonzalez-Cortazar M, Tortoriello J. Anxiolytic and antidepressant-like activity of a standardized extract from Galphimia glauca. Phytomedicine. 2006 Jan;13(1-2):23-8. doi: 10.1016/j.phymed.2005.03.003. Epub 2005 Jun 28. PMID 16360929
- [Result] Herrera-Ruiz M, Gonzalez-Cortazar M, Jimenez-Ferrer E, Zamilpa A, Alvarez L, Ramirez G, Tortoriello J. Anxiolytic effect of natural galphimines from Galphimia glauca and their chemical derivatives. J Nat Prod. 2006 Jan;69(1):59-61. doi: 10.1021/np050305x. PMID 16441069
- [Result] Mangas S, Bonfill M, Osuna L, Moyano E, Tortoriello J, Cusido RM, Pinol MT, Palazon J. The effect of methyl jasmonate on triterpene and sterol metabolisms of Centella asiatica, Ruscus aculeatus and Galphimia glauca cultured plants. Phytochemistry. 2006 Sep;67(18):2041-9. doi: 10.1016/j.phytochem.2006.06.025. Epub 2006 Jul 28. PMID 16876832
- [Result] Aguilar-Santamaria L, Ramirez G, Herrera-Arellano A, Zamilpa A, Jimenez JE, Alonso-Cortes D, Cortes-Gutierrez EI, Ledesma N, Tortoriello J. Toxicological and cytotoxic evaluation of standardized extracts of Galphimia glauca. J Ethnopharmacol. 2007 Jan 3;109(1):35-40. doi: 10.1016/j.jep.2006.06.013. Epub 2006 Jul 8. PMID 16930894
- [Result] Herrera-Arellano A, Jimenez-Ferrer E, Zamilpa A, Morales-Valdez M, Garcia-Valencia CE, Tortoriello J. Efficacy and tolerability of a standardized herbal product from Galphimia glauca on generalized anxiety disorder. A randomized, double-blind clinical trial controlled with lorazepam. Planta Med. 2007 Jul;73(8):713-7. doi: 10.1055/s-2007-981539. Epub 2007 Jun 11. PMID 17562493
- [Result] Osuna L, Moyano E, Mangas S, Bonfill M, Cusido RM, Pinol MT, Zamilpa A, Tortoriello J, Palazon J. Immobilization of Galphimia glauca plant cell suspensions for the production of enhanced amounts of Galphimine-B. Planta Med. 2008 Jan;74(1):94-9. doi: 10.1055/s-2007-993763. Epub 2008 Jan 4. PMID 18176908
- [Result] Jimenez-Ferrer E, Herrera-Ruiz M, Ramirez-Garcia R, Herrera-Arellano A, Tortoriello J. Interaction of the natural anxiolytic Galphimine-B with serotonergic drugs on dorsal hippocampus in rats. J Ethnopharmacol. 2011 Sep 1;137(1):724-9. doi: 10.1016/j.jep.2011.06.029. Epub 2011 Jul 1. PMID 21742023
- [Result] Herrera-Arellano A, Jimenez-Ferrer JE, Zamilpa A, Garcia-Alonso G, Herrera-Alvarez S, Tortoriello J. Therapeutic effectiveness of Galphimia glauca vs. lorazepam in generalized anxiety disorder. A controlled 15-week clinical trial. Planta Med. 2012 Sep;78(14):1529-35. doi: 10.1055/s-0032-1315110. Epub 2012 Jul 24. PMID 22828921
- [Result] Gonzalez-Cortazar M, Herrera-Ruiz M, Zamilpa A, Jimenez-Ferrer E, Marquina S, Alvarez L, Tortoriello J. Anti-inflammatory activity and chemical profile of Galphimia glauca. Planta Med. 2014 Jan;80(1):90-6. doi: 10.1055/s-0033-1360150. Epub 2013 Dec 11. PMID 24338551
- [Result] Abarca Vargas R, Zamilpa A, Aguilar FA, Herrera-Ruiz M, Tortoriello J, Jimenez-Ferrer E. Pharmacokinetic study in mice of galphimine-A, an anxiolytic compound from Galphimia glauca. Molecules. 2014 Mar 12;19(3):3120-34. doi: 10.3390/molecules19033120. PMID 24625685
- [Result] Jimenez-Ferrer E, Santillan-Urquiza MA, Alegria-Herrera E, Zamilpa A, Nogueron-Merino C, Tortoriello J, Navarro-Garcia V, Aviles-Flores M, Fuentes-Mata M, Herrera-Ruiz M. Anxiolytic effect of fatty acids and terpenes fraction from Aloysia triphylla: Serotoninergic, GABAergic and glutamatergic implications. Biomed Pharmacother. 2017 Dec;96:320-327. doi: 10.1016/j.biopha.2017.10.024. Epub 2017 Oct 7. PMID 29017144
- [Result] Santillan-Urquiza MA, Herrera-Ruiz M, Zamilpa A, Jimenez-Ferrer E, Roman-Ramos R, Tortoriello J. Pharmacological interaction of Galphimia glauca extract and natural galphimines with Ketamine and Haloperidol on different behavioral tests. Biomed Pharmacother. 2018 Jul;103:879-888. doi: 10.1016/j.biopha.2018.04.082. Epub 2018 Apr 24. PMID 29710504
- [Derived] Romero-Cerecero O, Islas-Garduno AL, Zamilpa A, Herrera-Arellano A, Jimenez-Ferrer E, Tortoriello J. Galphimine-B Standardized Extract versus Alprazolam in Patients with Generalized Anxiety Disorder: A Ten-Week, Double-Blind, Randomized Clinical Trial. Biomed Res Int. 2019 Jan 30;2019:1037036. doi: 10.1155/2019/1037036. eCollection 2019. PMID 30834253